CLINICAL TRIAL: NCT00901082
Title: The Effectiveness of Information and Relaxation on Pre-procedural Block Anxiety and Procedural Discomfort During Medial Branch Block: a Randomized Controlled Trial
Brief Title: The Effectiveness of Information and Relaxation on Pre-procedural Block Anxiety and Procedural Discomfort During Medial Branch Block
Acronym: TIRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louise Lamb (Other)
Responsible Party: Sponsor-Investigator, Louise Lamb, Nurse, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GEN08-051
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Pain
Keywords: chronic pain; anxiety; intervention; information; relaxation
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- information and relaxation (Active Comparator): will receive the intervention that consist of information and relaxation
  Interventions: Behavioral: Relaxation and information session
- No intervention (No Intervention): No specific intervention before the medial branch block.

INTERVENTIONS:
Behavioral: Relaxation and information session — Relaxation and information session before the medial branch block
  Arms: information and relaxation

SUMMARY:
Patient presenting to chronic pain clinics frequently undergo diagnostic and therapeutic spinal injections as part of their treatment. These procedures can cause significant level of apprehension in patients, which can lead to increased procedural times, increased procedural pain and reluctance to continue with the treatment program. It appears that certain interventions could reduce the anxiety and catastrophization levels and modify pain perception during medical procedures. The investigators therefore sought to evaluate the effect of a single 30 minutes information session which includes relaxation training administered 5 to 6 days before the nerve block procedure on patient's anxiety and catastrophization levels prior to the procedure and pain scores during the procedure, as well as the overall level of satisfaction with care received.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled to have a medial branch block
* over 18 years of age

Exclusion Criteria:

* adult able to give their own consent
* patients who had a previous nerve block
* patients who have a major psychiatric illness
* patients who do not understand English or French

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in the anxiety level prior to the nerve block as per the state trait anxiety questionnaire | 5-7 days (Second visit and Day of block)

SECONDARY OUTCOMES:
Perceived pain as measured by NRS (numerical rating scale) | Throughout the study (Baseline, day of block and 1 month after)
Unchanged catastrophization level | Baseline and day of block
Satisfaction level of the overall experience | Day after the block
Ease of performing the nerve block | Day of block

CONTACTS AND LOCATIONS:
Locations (1):
- MUHC, Montreal General Hospital, Montreal, Quebec, Canada